CLINICAL TRIAL: NCT00232193
Title: Steroid Adjunctive Treatment at Initiation of Avonex Therapy for Patients With Mono-Symptomatic or Relapsing-Remitting Multiple Sclerosis
Brief Title: Safety/Effectiveness of Adding Monthly Dexamethasone to Weekly Avonex for MS
Status: Completed | Type: Observational
Sponsor: Providence Multiple Sclerosis Center (Other)
Collaborators: Biogen (Industry)
Responsible Party: Stanley Cohan, MD, Medical Director, Providence MS Center
Other Study IDs: 011-03-AVX
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Relapsing-remitting Multiple Sclerosis; Clinically Isolated Syndrome
Keywords: Multiple Sclerosis; Interferon Beta 1-a; Pulsed steroids
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IFNβ+DS group: IFNβ+DS group received lyophilized Avonex 30mcg IM weekly plus dexamethasone 160 mg IV every 4 weeks for 52 weeks and was treated with Avonex 30mcg IM weekly from week 53 to 104
- IFNβ group: IFNβ group received lyophilized Avonex 30mcg IM weekly for 104 weeks

SUMMARY:
The purpose of the study is to determine whether giving intravenous dexamethasone every 4 weeks during the first 12 months of weekly Avonex dosing will reduce the progression of functional impairment, brain atrophy, relapse rate and frequency, and new and enlarging brain lesions over the first 24 months of Avonex therapy in patients with relapsing-remitting or mono-symptomatic multiple sclerosis.

DETAILED DESCRIPTION:
Beta Interferon-1a (Avonex)was approved by the FDA in 1996 to treat relapsing-remitting multiple sclerosis. Clinical trials have shown evidence in the reduction of relapses and progression of neurological and cognitive disability with the use of Avonex, as well as reduction in brain atrophy and new MS lesions on MRI were observed. Despite this, Avonex does not abolish disease activity, therefore, there is frequent need for adjunctive therapy, such as short courses of corticosteroids.

This study will research the value of adding monthly pulsed corticosteroids as adjunctive therapy during the first year of Avonex use to determine: a)safety and tolerability b)if this therapy will reduce the progression of functional impairment, and c)if this therapy will reduce the progression of whole brain atrophy over a 13 month observation period.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients between the ages of 18-55 years inclusive
* have provided informed consent to be screened for the study
* have been diagnoses as having MS
* meet the McDonald diagnostic criteria for RRMS or CHAMPS criteria for CIS
* have an EDSS score of 0.0-3.5
* have had no immunomodulator or cytoxic agents and have had no steroids or other immunosuppressants within 30 days prior to Baseline Visit
* must have had a brain MRI scan demonstrating lesions consistent with MS on T2-weighted or FLAIR images
* subjects must be willing and able to participate in all aspects of the study, including use of study medications as prescribed, and screening and follow-up clinical and MRI assessments

Exclusion Criteria:

* type I of type II diabetes
* uncontrolled hypertension (systolic >160 or diastolic >100 despite medication therapy)
* history of suicidal ideation
* history of psychosis
* history of alcoholism or other substance abuse
* clinically significant coronary artery disease
* history of hepatic failure and chronic renal failure
* history of cancer other than basal or squamous cell carcinoma of the skin
* pregnancy or unwillingness to use adequate precautions to prevent pregnancy during the duration of this study
* nursing mothers
* history of stroke, dementia, seizure disorder, peripheral neuropathy, Parkinsonism, myasthenia, myelopathy or other primary degenerative disease of the central or peripheral nervous system
* history of peptic ulcer disease
* history of intolerance to corticosteroids or allergy to albumin
* history of osteoporosis
* history of Lupus, Sjogrens syndrome, Lyme disease or syphilis
* abnormal laboratory results indicative of significant hepatic, renal, hematopoetic, or coagulation dysfunction
* the entity of any disease entity, which in the opinion of the investigators would potentially prevent the patient from successfully completing 2 years participation in this trial or confound the observations made during this trial
* prior use of Avonex, Betaseron, Rebif, mitoxantrone, cyclophosphamide, azothioprine, methotrexate, cladribine, cyclosporin, CellCept, IVIG, natalizumab, anti T-cell or anti B-cell antibodies, plasmapheresis or other systemic immunosuppressant or cancer chemotherapeutic agents
* unwillingness or inability to comply with all the requirements of the protocol
* known diagnosis of osteoporosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Treatment-naive MS patients with either RRMS or CIS, of either gender, between 18 to 55 years of age inclusive, with baseline EDSS of 0 to 3.5, fulfilling McDonald criteria for MS or CHAMPS criteria for CIS, were randomly assigned to one of two treatment groups.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2003-12; Primary Completion 2008-12 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley L. Cohan, M.D., Ph.D., Principal Investigator — Providence Multiple Sclerosis Center
Locations (1):
- Providence MS Center, Portland, Oregon, United States